CLINICAL TRIAL: NCT06880081
Title: A Phase 1b, Open-label, Single-arm, Dose-escalation Study of PN20 in Patients with Primary Immune Thrombocytopenia (ITP)
Brief Title: Study of PN20 in Adult Patients with Primary Immune Thrombocytopenia (ITP)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Peg-Bio Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQPJ-PN20-ITP-Ib
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
Keywords: Primary Immune Thrombocytopenia (ITP); thrombopoietin receptor agonist; PN20
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PN20 treatment group-single dose (Experimental): A single dose of PN20 will be administered.
  Interventions: Drug: PN20 treatment

INTERVENTIONS:
Drug: PN20 treatment — Three dose cohorts, single dose, subcutaneous injections
  Other Names: thrombopoietin receptor agonist

SUMMARY:
The main aim of this clinical trial is to assess the safety and tolerability of PN20 in adult patients with primary immune thrombocytopenia (ITP). The main questions it aims to answer are:

* Is PN20 safe in these patients?
* Could these patients potentially benefit from PN20 treatment?

Participants will

* Receive one subcutaneous injection of PN20 according to weight;
* Visit the clinic for assessment.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm, dose-escalation Phase1b study aimed at evaluating the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), immunogenicity, and preliminary efficacy of a single dose of PN20 in adult patients with primary immune thrombocytopenia (ITP).

The trial is a dose escalation study, including Screening (no more than 14 days), Treatment (single dose) and the post-treatment follow-up (4 weeks).

And the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary efficacy of PN20 in ITP will be assessed in this study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Aged between 18 and 65 years (inclusive), male or female;
2. Diagnosed with primary immune thrombocytopenia (ITP) and have a disease course of more than 6 months;
3. Patients who have no response or relapsed after splenectomy. Or patients who have not been splenectomised and have completed at least 1 prior treatment for ITP (such as glucocorticoids, immunoglobulin) and have failed to respond or relapsed after treatment;
4. During screening period, the mean of two platelet counts must be < 30 × 10^9/L, with none >35 × 10^9/L;
5. Fully understand and are able to comply with the requirements of the protocol, voluntarily participate and sign the informed consent form.

Key Exclusion Criteria:

1. History of bone marrow stem cell disorder. Any abnormal bone marrow findings other than typical of ITP.
2. Any active malignancy. If prior history of cancer other than basal cell carcinoma or cervical carcinoma in situ, no treatment or active disease within 5 years prior to signing the ICF.
3. Diagnosed with arterial thrombotic disease (such as cerebral thrombosis, transient ischemic attack, myocardial infarction, peripheral arterial disease, etc.); Patients with a history or complications of venous thrombosis (such as deep vein thrombosis, pulmonary embolism); or patients who are using anticoagulants or antiplatelet drugs at the beginning of screening.
4. Subjects who have used romiplostim or its analogs in the past and have not responded.
5. Subjects who have used eltrombopag, haitubopag, avatubopag, recombinant human thrombopoietin (rhTPO), or other drugs with c-MPl stimulating effects within the 4 weeks prior to signing the ICF.
6. Received any anti-malignancy agents (e.g., cyclophosphamide, mercaptopurine, vincristine, vinblastine, interferon-alfa) within 8 weeks prior to signing the ICF.
7. Less than 4 weeks since end of any clinical trials about therapeutic drug or device prior to signing the ICF.
8. Laboratory abnormalities with clinical significance at screening visit.
9. In the opinions of investigators, the patients are not suitable for participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE) | Treatment and post-treatment follow-up period (28 days after a single dose)
  The incidence of adverse events related to PN20.

SECONDARY OUTCOMES:
The percentage of subjects who reach the target therapeutic platelet level after administration | Treatment and post-treatment follow-up period (28 days after a single dose)
  It is defined as the proportion of subjects whose platelet count reaches at least 2 times the baseline platelet count within 28 days after administration and is within the range of 50×10^9/L to 450×10^9/L (inclusive).

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Principal Investigator — Chinese Academy of Medical Sciences
Locations (5):
- China (5):
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jining First People's Hospital, Jining, Shandong
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No